CLINICAL TRIAL: NCT06797687
Title: Mitral Valve Annulus Assessment, a Comparison Between 3D-TOE, CCT and Surgical Ring
Brief Title: Mitral Valve Annulus Assessment, Multimodality Imaging
Acronym: MAS-3D
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7065
Record Dates: First submitted 2025-01-23; First posted 2025-01-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-01

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac computed tomography — Mitral valve annulus measurements in the enrolled patients obtained will be obtained from: coronary CT scan, intraoperative transesophageal echocardiography and the ring surgically implanted during surgery.
  Other Names: Three-dimensional transesophageal echocardiography; Mitral valve surgical repair

SUMMARY:
The success of mitral valve repair with annuloplasty depends on the repair technique and on the choice of a ring with appropriate dimensions related to mitral annulus. Intraoperatively, the choice of the prosthetic ring size is made by the surgeon using special gauges that are placed on the anterior mitral leaflet (having the trigons and commissures as anatomical findings), a method considered the gold standard for defining annulus size. However, it is performed in cardioplegia, without considering annulus shape and motion during cardiac cycle. Three-dimensional techniques are fundamental in evaluating mitral valve structure and its changes during cardiac cycle; three-dimensional transoesophageal echocardiography (3D-TOE) has been proven to be essential for the anatomo-functional characterization of mitral valve apparatus in patients undergoing surgically mitral valve repair. It also allows the measurement of quantitative parameters useful in determining the size of the annuloplasty ring, such as A2 scallop height, intertrigonal distance, intercommissural diameter and total annular perimeter size, that will support the surgeon's choice on the dimensions of the ring to be implanted. Cardiac computed tomography (CCT) plays a key role for device sizing in patients undergoing transcatheter mitral valve replacement; it provides isotropic sub-millimetre spatial resolution and it is the gold standard for geometric characterisation of the mitral valve and for assessment of the spatial relationship of mitral valve apparatus to adjacent anatomical structures. In patients undergoing mitral valve surgery it is foremost performed to exclude coronary artery disease, as stated by European Society of Cardiology (ESC) guidelines. Several studies have compared CCT with 3D-TOE in sizing the mitral valve apparatus: Shanks et al. have demonstrated a good correlation between the two techniques in measuring intercommissural diameter; Hirasawa et al. have demonstrated a good correlation in evaluating intertrigonal distance. Only one study has compared the measures of the annulus obtained by CCT with the prosthetic ring (Alkhadi et al.) and only for 9 patients the intercommissural diameter was compared to the prosthetic ring, obtaining a good correlation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with severe mitral valve regurgitation, with an indication for surgical treatment of the valvopathy and who have undergone cardiac surgery for mitral valve surgery with prosthetic ring implantation
* Pre-operative coronary CT scan as a diagnostic tool for the exclusion of coronary artery disease (in accordance with the guidelines for chronic coronary syndrome and valvulopathy) with adequate image quality to allow measurement of the mitral annulus
* Availability of adequate three-dimensional echocardiographic reconstructions of the mitral valve apparatus at the intraoperative transesophageal echocardiogram to allow measurements of the annulus
* Provision of informed consent prior to enrolment

Exclusion Criteria:

* Implantation of mitral valve prosthesis due to inability to perform mitral valve repair
* Unavailability of CCT scan
* Unavailability of intraoperative transesophageal echocardiogram
* Unavailability of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe mitral regurgitation with indication to surgical treatment who are elegible according to inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Comparison between 3D-TOE and CCT | 48 hours
  The reliability of mitral annulus measurements obtained by three-dimensional transesophageal echocardiography (evaluated in terms of anterior leaflet length, intertrigonal distance and intercommissural diameter) compared to cardiac computed tomography.

SECONDARY OUTCOMES:
Comparison between CCT and surgery | 48 hours
  The reliability of mitral annulus measurements obtained by cardiac computed tomography with the dimensions of the implanted ring during cardiac mitral valve repair surgery.
Comparison between 3D-TOE and surgery | 24 hours
  The reliability of mitral annulus measurements obtained by intraoperative three-dimensional transesophageal echocardiogram with the dimensions of the implanted ring during cardiac mitral valve repair surgery
Determination of the best measure | 1 year
  To demonstrate whether any of the individual variables (anterior leaflet height, intertrigonal distance and intercommissural diameter) correlates better with the size of the implanted ring size (from the available data, the intercommissural diameter has shown a better correlation than the intertrigonal distance, although there are no studies that have directly compared the two values).

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Pasquini, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Cardiologia, Roma, Italy